CLINICAL TRIAL: NCT04563143
Title: Novel Paradigms of Deep Brain Stimulation for Movement Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Farmer Foundation (Unknown)
Responsible Party: Principal Investigator, Kenneth Baker, PhD, Co-Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1637
Record Dates: First submitted 2020-04-22; First posted 2020-09-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: deep brain stimulation; sensorimotor function; cognition
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Novel stimulation (Other): All subjects will undergo periods of stimulation using novel stimulation patterns
  Interventions: Other: Novel DBS Stimulation

INTERVENTIONS:
Other: Novel DBS Stimulation — Stimulation patterns will vary from the standard therapeutic approach in terms of frequency, contact location, and/or temporal pattern.

SUMMARY:
Investigators will enroll patients who are already selected to undergo deep brain stimulation surgery based on standard of care. The surgical implantation of the leads will be based on standard of care and will be completed with FDA-approved leads that are routinely used at Cleveland Clinic. The pulse generators (i.e. the battery) will also be standard. The research will characterize spontaneous and task-related changes in brain activity recorded from these regions alone and in relation to novel paradigms / settings of stimulation to learn how such paradigms impact both the symptoms of patients with Parkinson's disease and the underlying neural activity of the target brain region. Of particular interest is to learn if the novel paradigms of stimulation will have a lower impact on cognitive function than current settings of stimulation.To date, current DBS settings are continuous. That is, stimulation runs at approximately 200 pulses per second, all day long, day and night.

The novel settings that investigators will study are part of a translational pipeline at Cleveland Clinic. Dr. Ken Baker and Dr. Machado are partners in the lab and in clinical research. Dr. Baker has completed preclinical research that has shown that it is possible to achieve excellent relief of parkinsonian symptoms with intermittent types of stimulation known as coordinated reset. In other words, Dr Baker found that using a lower dose of stimulation in an intermittent fashion can maintain the same level of symptom control. Furthermore, a lower dose of stimulation could have less effects on cognitive symptoms.

In order to test these novel paradigms of stimulation, investigators will study patients immediately after DBS and over time. The immediate research will be done starting on the third day after implantation of the DBS lead(s), having the systems externalized for nine days. The long-term research will be conducted with patients already fully implanted and healed from surgery. In addition to evaluating for motor and cognitive tasks using computer based assessments, investigators will utilize non-invasive electrophysiological measures including EEG, EMG, MEG, and wearable accelerometer/gyroscopes to better characterize the effects of stimulation settings.

DETAILED DESCRIPTION:
The experimental design will include procedures to address each specific aim, with most involving a within-subjects approach that examines the effect of different levels of treatment (e.g., no therapy, traditional DBS, novel DBS) on neurological function, including dependent variables derived from tests of motor and cognitive function. This approach will extend to the electrophysiological data as well; where the relative effect of each level of treatment on spontaneous- (e.g., resting beta and gamma band power) and task-related (i.e., evoked or event-related potential latency and amplitude characteristics) cerebral rhythms will be quantified for each subject and further aggregated to characterize group-level effects (see data analysis below).

Prior to surgery, participants will undergo additional brain imaging procedures in order to characterize the anatomical and functional connectivity of the brain region to be targeted during surgical lead placement and the cerebral cortex. The additional imaging sets will include DTI and resting state functional MRI scans that will add an additional 30-45 minutes to the standard of care pre-operative clinical MR procedure.

Following standard of care placement of the DBS lead(s) within the targeted brain region, access to the lead for study-related activities will be achieved by attaching a disposable extension to the end of the lead that is lodged subcutaneously, extracranially. The disposable extension will then be tunneled to a site remote to that of the surgery in order to minimize risk of contamination of the permanently implanted hardware. The recording equipment will then be connected to the externalized extension, thus enabling study-related DBS delivery and the recording of local field potentials (LFP) from the targeted brain region.

Study-related activities will start the third morning after DBS surgery to allow the patient time to recover from the implant procedure (start may be delayed if additional recovery is deemed warranted through consultation with clinical care team). It is expected that the study testing will continue through post-implant day 9, with the second standard of care DBS implant surgery performed on post-implant day 10. During the externalization period, subjects will participate in daily data collection tasks for up to 8 hours per day, with study-related activities performed in short segments, broken up across morning and afternoon sessions. Once testing is completed in the operationally-defined medication OFF state, patients will be permitted to take their usual dose of medication and testing will continue. Frequent rest periods will be included within each testing block to minimize fatigue effects and improve data quality. Electrophysiological recordings may also be performed when the patient is not in the laboratory, including overnight during sleep, using portable recording equipment and activity monitors that resemble a holster device. Recordings will be made using either a commercially-available cap electrode system that is placed temporarily during each experimental session or using standard cup electrodes affixed to the scalp using either standard methods (i.e., collodion or electrode paste). If collodion electrodes are used, collodion electrodes will remain on the patient for several days in a row up to the duration of the externalization period. Daily checks will be performed to ensure the integrity of the electrode interface and electrodes will be re-gelled or re-applied as needed.

Daily study-related activities within the laboratory will include 1) spontaneous recordings made with the patient at rest, 2) motor and cognitive task-synchronized recordings, and 3) somatosensory evoked potentials, and 4) evoked potentials elicited by direct stimulation of the deep brain target region. On the first day of testing, a monopolar threshold review, similar to what is performed as part of standard of care clinical DBS programming may be performed. This involves careful titration of the settings of electrical stimulation delivered via the DBS lead in order to determine thresholds for sensorimotor and other side-effects and will help to set the upper limits of stimulation delivered as part of the experimental procedures. Moreover, this process will be used to characterize the therapeutic benefits derived from DBS. In all cases, stimulation will be limited to less than the approved charge density safety limit of 30 microcoulombs/cm2 per phase. On certain days, patients may be asked to arrive to the test location after an overnight fast from their anti-PD medications in order to characterize the effect of dopaminergic medications on experimental responses. Finally, daily schedules may be altered based upon patient fatigue as well as potential scheduling conflicts (e.g., MRI or MEG availability) and the total number of days the patient is externalized may be shortened at the discretion of the surgical team, including the need to accommodate operating room scheduling.

A minimum of six months after surgery, participants will be asked to return for a follow-up, approximately 4-hour research visit to evaluate therapeutic outcomes. Specifically, patients will be asked to return to the main campus laboratory after an overnight fast from their anti-parkinsonian medications. During that visit, the efficacy of the patient's standard-of-care DBS programming settings (i.e., the settings set by their treating physician as part of their routine, post-op clinical care) will be evaluated through blinded scoring using subscales of the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic Parkinson's disease for greater than 3 years
* determined appropriate for deep brain stimulation surgery
* able to give consent

Exclusion Criteria:

* secondary Parkinson's disease, stroke, progressive central nervous system disease
* dementia that disallows the subject ability to consent
* current alcohol or substance abuse
* hearing or visual impairment precluding cognitive or sensory testing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Upper extremity motor speed | Post operative externalization days 1 through 9
  Patients will complete arm movements in response to cues presented on a computer. The speed of movements will be compared between novel and therapeutic stimulation
Verbal Fluency | Post operative externalization days 1 through 9
  Change in the number words that patients generate to letter or semantic category cues will be compared between novel and therapeutic stimulation

SECONDARY OUTCOMES:
Cognitive Reaction Time | Post operative externalization days 1 through 9
  Subjects will complete one or more measures of cognitive processing requiring speeded responses to stimuli. Changes in reaction time will be compared between novel and therapeutic stimulation
EEG - sensorimotor evoked potentials | Post operative externalization days 1 through 9
  Sensory and motor-locked activity at scalp and deep brain stimulation electrodes will be compared between novel and therapeutic stimulation
EEG - Oscillatory activity | Post operative externalization days 1 through 9
  Power in standard frequency bands at both scalp and DBS electrodes will be examined with the patient at rest and compared between novel and therapeutic stimulation
EMG | Post operative externalization days 1 through 9
  Electromyography will be recorded in response to active and passive movement and latency and amplitude will be compared between novel and therapeutic stimulation
fMRI - Bold response | Post operative externalization days 1 through 9
  Pattern of fMRI activity will be compared between novel and therapeutic stimulation
MEG | Post operative externalization days 1 through 9
  Pattern of magnetoencephalogram activity will be compared between novel and therapeutic stimulation
Movement Disorders Society Unified Parkinson Disease Rating Scale - III | 6 months after DBS surgery
  Gold standard clinician rating scale of Parkinson's symptoms will be compared between novel and therapeutic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Baker, PhD, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States